CLINICAL TRIAL: NCT05013177
Title: Effect of COVID-19 Vaccine on Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kelvin KF Tsoi, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2021.448
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Blood Pressure; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate (1) if COVID-19 vaccine impacts on blood pressure, (2) the extent of impact on blood pressure (if any), and (3) which groups of subjects are more susceptible to be affected by COVID-19 vaccine on blood

DETAILED DESCRIPTION:
Coronavirus disease 19 (COVID-19), which is caused by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), has elicited global pandemic since January 2020. Until the end of June 2021, the virus has caused 182 million confirmed COVID-19 cases and 3.95 million deaths worldwide. To stop the spread of virus, there has been rapid development of vaccine against SARS-CoV-2. Currently there has been 9 vaccines authorized for emergency use, and 8 vaccines received full approval for use in various countries. Extensive studies have been showing the efficacy of different types of vaccines against COVID-19 and its variants. Safety of COVID-19 vaccines has been a concern. Despite safety profile of different vaccines demonstrated in phase 2/3 trials, there has been evolving evidence on adverse effects of some particular COVID-19 vaccines. One of the mostly known example is vaccine-induced thrombotic thrombocytopenia (VITT). Case series report4 and observational studies on ChAdOx1 nCoV-19 vaccine showed high level of autoantibodies to platelet factor-4 (PF4) which could contribute to microvascular damage, micro-bleeding and platelet activation and therefore causes event of thrombosis. Apart from the thrombotic risk of ChAdOx1 nCoV-19 vaccine, there has been studies providing the preliminary data on effect of mRNA-based COVID-19 vaccine on blood pressure. Yet there remains lack of evidence and detailed description on effect of COVID-19 vaccines and blood pressure along the time. Given the vast population of hypertensive patients worldwide, the increasing number of people being vaccinated and the importance of blood pressure level to various human organs, it is essential to investigate the short- and long-term effect of COVID-19 vaccine on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years old or above
* Subjects with home blood pressure monitoring device
* Subjects with smartphone and with HealthCap application downloaded
* Subjects who understand Chinese to make an informed consent

Exclusion Criteria:

* Subjects unable to take regular home blood pressure measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants attending CUHK Medical Centre community vaccination centre or CUHK Medical Clinic to receive COVID-19 vaccination will be invited to the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
To investigate if COVID-19 vaccine impacts on blood pressure. | 6 weeks
  To measure blood pressure at the time of COVID-19 vaccination and during follow-up